CLINICAL TRIAL: NCT01229033
Title: Ablating Atrial Tachycardias Occuring During Ablation of Complex Fractionated Electrograms in Persistent AF - ATTAC CFAE Trial
Brief Title: Ablating Atrial Tachycardias Occuring During Ablation of Complex Fractionated Electrograms in Persistent AF
Acronym: ATTAC CFAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Klinik für Kardiologie, Klinikum Karlsruhe, Prof. Dr. C. Schmitt (Unknown)
Responsible Party: Isabel Deisenhofer, MD and Clemens Jilek, MD, Deutsches Herzzentrum München
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-001
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation; Ablation; Atrial Flutter
Keywords: Atrial fibrillation; ablation; atrial flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Electric Countershock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablation (Active Comparator): Ablation of atrial tachycardia
  Interventions: Procedure: Ablation
- Cardioversion (Active Comparator): Cardioversion of atrial tachycardia
  Interventions: Procedure: Cardioversion

INTERVENTIONS:
Procedure: Ablation — Ablation of atrial tachycardia
  Arms: Ablation
Procedure: Cardioversion — Cardioversion of atrial tachycardia
  Arms: Cardioversion

SUMMARY:
Catheter ablation has proven to be an effective treatment option in patients suffering from symptomatic persistent atrial fibrillation (AF). Catheter ablation consists of two major steps: (1) Isolation of pulmonary veins to abolish the trigger of atrial fibrillation and (2) modification of left atrial and eventually right atrial substrate by ablation of complex fractionated atrial electrograms (CFAE). CFAE are mainly found at the ostia of the pulmonary veins, around the left atrial appendage, at the mitral annulus and the septum.

When ablating CFAE 40-65% of the patients show a regularization of AF to an atrial tachycardia (AT) that can be macro- or micro-reentrant (localized re-entry). Until now the significance of the AT is unclear.

In the following study we examine the hypothesis that an ablation of AT occuring during CFAE ablation (group 1) significantly improves outcome defined as freedom of atrial arrhythmia (AF or AT) compared to patients that are cardioverted when AF has regularized to AT (group 2).

ELIGIBILITY:
Inclusion Criteria:

* Patients (>=18 und < 80 years) with symptomatic persistent AF (AF episode enduring at least 7 days) but are successfully convertable in sinus rhythm (SR).
* At least one unsuccessful attempt of antiarrhythmic drug (betablocker or class I oder III).
* Oral anticoagulation with phenprocoumone or warfarine for at least 4 weeks prior to ablation with weekly documented INR > 2..
* Withdrawal of antiarrhythmic drugs at least 3 half times prior to ablation except amiodarone.
* Atrial tachycardia occurring during ablation of CFAE (defined as CL > 200 msec und stable activation sequence).

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial tachyarrhythmia
  Documented freedom from atrial tachyarrhythmia (AF or AT) during follow-up after first ablation.

SECONDARY OUTCOMES:
Procedural and safety data
  1. Duration of left atrial procedure, time of ablation, time of radiation and radiation dose from randomization until the end of the procedure.
  2. In case of recurrence, characteristic of predominant tachyarrhythmia (AF or AT).
  3. Safety parameters (pericardial tamponade, thrombembolic complications).
  4. Number of re-ablations.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Deisenhofer, MD, Study Chair — Deutsches Herzzentrum München; Clemens Jilek, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (2):
- Germany (2):
  - Klinikum Karlsruhe, Karlsruhe
  - Deutsches Herzzentrum München, München